CLINICAL TRIAL: NCT04376827
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Guselkumab in Subjects With Active Lupus Nephritis
Brief Title: A Study of Guselkumab in Participants With Active Lupus Nephritis
Acronym: ORCHID-LN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges, J&J Innovative Medicine decided to stop screening and terminate the study early. This decision was not based on a safety concern.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108766; 2018-003155-38 (EudraCT Number); CNTO1959LUN2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Guselkumab+Standard of Care (Experimental): Participants will receive guselkumab Dose 1 intravenously (IV) at Weeks 0, 4 and 8 and guselkumab Dose 2 subcutaneous (SC) every 4 weeks (q4w) from Week 12 through Week 48 along with standard-of-care treatment of mycophenolate mofetil (MMF)/mycophenolic acid (MPA) and glucocorticoids. Participants who achieved complete renal response (CRR) at Week 48 and 52 and have completed the Week 52 assessment may have the option to participate in the long-term extension (LTE).
  Interventions: Drug: Guselkumab Dose 1; Drug: Guselkumab Dose 2; Drug: Standard-of-care treatment
- Placebo+Standard of Care (Placebo Comparator): Participants will receive placebo IV at Weeks 0, 4 and 8 and placebo SC q4w from Week 12 through Week 48 along with standard-of-care treatment of MMF/MPA and glucocorticoids. Participants who achieved complete renal response (CRR) at Week 48 and 52 and have completed the Week 52 assessment may have the option to participate in the LTE of the study.
  Interventions: Drug: Placebo; Drug: Standard-of-care treatment

INTERVENTIONS:
Drug: Guselkumab Dose 1 — Participants will receive guselkumab Dose 1 via IV administration.
  Other Names: CNTO 1959
  Arms: Guselkumab+Standard of Care
Drug: Placebo — Participants will receive placebo IV at Weeks 0, 4 and 8 (that is, 3 IV doses) and placebo SC q4w from Week 12 through Week 48.
  Arms: Placebo+Standard of Care
Drug: Guselkumab Dose 2 — Participants will receive guselkumab Dose 2 via SC route.
  Other Names: CNTO1959
  Arms: Guselkumab+Standard of Care
Drug: Standard-of-care treatment — Participants will receive standard of care treatment including MMF/MPA and glucocorticoids from Week 12 through Week 48.

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab in participants with active lupus nephritis (LN).

DETAILED DESCRIPTION:
Guselkumab is a monoclonal antibody (mAb) that binds to human interleukin (IL)-23 with high affinity and blocks binding of extracellular IL-23 to cell surface IL-23 receptor, inhibiting IL 23 specific intracellular signaling and subsequent activation and cytokine production. It is used in treatment of plaque psoriasis, psoriatic arthritis, generalized pustular psoriasis, erythrodermic psoriasis. Lupus is a heterogeneous autoimmune disease with lesions confined to skin (cutaneous lupus erythematosus [CLE]) to others that involve 1 or more vital internal organs (systemic lupus erythematosus [SLE]). Renal involvement due to SLE is termed lupus nephritis (LN). There is a high unmet need for new treatment options in LN that are safe and effective, especially new therapies that can provide improved long-term efficacy over currently available therapies. This study will evaluate safety and efficacy of guselkumab added to standard-of-care compared to placebo added to standard-of-care. Total duration of study is up to 68 weeks: a less than or equal to 8 week screening period, a 48 week double-blind treatment period, a 12 week safety follow-up period after last dose. Participants who complete the assessments at Week 52 and have achieved complete renal response (CRR) may have the option to participate in the long-term extension (LTE) of study through Week 152 and the 12-week safety follow-up visit. Hypothesis of this study is that guselkumab plus standard-of-care is superior to placebo plus standard-of-care in participants with active LN as measured by the proportion of participants inducing at least a 50 percentage reduction of proteinuria with protocol specified steroid tapering regimen at Week 24. Safety assessments include Adverse events (AEs), clinical laboratory tests (hematology and chemistry), systolic and diastolic blood pressures over time, monitoring for hypersensitivity reactions, AEs temporally associated with infusion, injection-site reactions, suicidality assessment, and early detection of active tuberculosis (TB).

ELIGIBILITY:
Inclusion Criteria:

* At screening and randomization, must be receiving oral glucocorticoids at minimum prednisone equivalent dose of 10 milligrams per day (mg/day) and maximum 1 mg/kg/day or less than or equal to (<=) 60 mg/day, whichever is lower. Treated for greater than or equal to (>=) 6 weeks with stable dosing >=2 weeks before randomization
* If receiving angiotensin-converting enzyme (ACE) inhibitor/angiotensin II receptor blockers (ARB), a stable dose for at least 2 weeks prior to randomization
* Positive antinuclear antibody (ANA; >= 1:80 titer by central laboratory test) or anti-double-stranded deoxyribonucleic acid (dsDNA) antibodies (>=30 international units per milliliter ([U/mL] by central laboratory test) detected at screening
* Kidney biopsy documentation of active International Society of Nephrology (ISN)/Renal Pathology Society (RPS) proliferative nephritis: Class III-IV (with or without class V membranous nephritis) within the last 6 months prior to screening or performed during screening
* Urine Protein to Creatinine Ratio (UPCR) >= 1.0 milligram/milligram (mg/mg) assessed on 2 first morning urine void specimens during screening. These 2 specimens do not need to be on consecutive days, however, 2 samples must be tested with UPCR >= 1.0 mg/mg in a row. The UPCR requirement must be met after at least 8 weeks of mycophenolate mofetil (MMF)/mycophenolic acid (MPA) treatment, and after stable glucocorticoid dosing is achieved at the dose intended at time of randomization

Exclusion Criteria:

* Comorbidities (other than lupus nephritis [LN], example, asthma, chronic obstructive pulmonary disease) which have required 3 or more courses of systemic glucocorticoids within the previous 12 months
* Has other inflammatory diseases that might confound the evaluations of efficacy, including but not limited to rheumatoid arthritis (RA), psoriatic arthritis (PsA), RA/lupus overlap, psoriasis, Crohn's disease, or active Lyme disease
* Received PO (orally) or intravenously (IV) cyclophosphamide within 3 months prior to randomization
* History of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, before screening
* History of being human immunodeficiency virus (HIV) antibody-positive, or tests positive for HIV at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (60):
- United States (8):
  - Medvin Clinical Research, Covina, California
  - UC San Diego, La Jolla, California
  - Academic Medical Research Institute, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Med Research, Inc., El Paso, Texas
- Argentina (8):
  - Centro Médico Reumatológico (OMI), Buenos Aires
  - Hospital Ramos Mejia, Caba
  - ARCIS Salud SRL Aprillus asistencia e investigacion, CABA
  - Instituto Medico Strusberg SA, Córdoba
  - Clinica Privada Velez Sarsfield, Córdoba
  - Instituto de Reumatologia - Ir Medical Center S.A., Mendoza
  - Instituto Médico de la Fundación de Estudios Clínicos (ECLIN), Rosario
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Mexico (6):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Centro de Investigacion y Tratamiento Reumatologico S C, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Unidad Reumatologica las Americas S.C.P., Mérida
  - Consultorio de Reumatologia, México
  - Unidad de Investigaciones Reumatologicas A.C, San Luis Potosí City
- Poland (3):
  - Uniwersyteckie Centrum Medyczne Klinika Nefrologii Transplantologii i Chorob Wewnetrznych, Gdansk
  - Uniwersytecki Szpital Kliniczny nr 1 im. N. Barlickiego, Lodz
  - Uniwersytecki Szpital Kliniczny we Wroclawiu, Wroclaw
- Russia (5):
  - LLL Medical Center Revma-Med, Kemerovo
  - Orenburg State Medical University, Orenburg
  - LLC Medical Sanitary Part No. 157, Saint Petersburg
  - LLC German Clinic, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
- Spain (8):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Fuenlabrada, Madrid
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Thailand (4):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai
  - Songklanagarind hospital, Hat Yai
- Ukraine (14):
  - Communal Noncommercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Municipal non-commercial enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - City Clinical Hospital No. 2, Kryvyi Rih
  - Medical Center 'Ok Clinic' of International Institute of Clinical Research LLC, Kyiv
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - Medical Center 'Consylium Medical', Kyiv
  - State Institution 'Institute of Nephrology of the National Academy of Medical Sciences of Ukraine', Kyiv
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - Multidisciplinary Medical Center of Odessa National Medical University, Odesa
  - Municipal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Ternopil
  - Medical Center LTD Health Clinic Department of Cardiology and Rheumatology, Vinnytsia
  - MNPE 'Vinnytsia Regional Clinical Hospital named after M.I. Pyrogov of Vinnytsia Regional Council', Vinnytsia
  - Medical Center LLC 'Modern Clinic', Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Anders HJ, Chan TM, Sanchez-Guerrero J, Wofsy D, Bensley K, Kim L, Lo KH, Shu C, Shao J, Karyekar CS, Diamond B. Efficacy and safety of guselkumab in patients with active lupus nephritis: results from a phase 2, randomized, placebo-controlled study. Rheumatology (Oxford). 2025 May 1;64(5):2731-2740. doi: 10.1093/rheumatology/keae647. PMID 39673415
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520
- See also: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Guselkumab in Subjects with Active Lupus Nephritis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108766&attachmentIdentifier=0153a0b8-08f3-4f41-a43e-b27e5d1f2be3&fileName=CR108766_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified by geographic region (North America, Latin America, Asia Pacific and Europe) and Urine Protein to Creatinine Ratio (UPCR) level (less than [<] 3 milligrams per milligram [mg/mg] and greater than or equal to [>=] 3 mg/mg).
Groups:
- Placebo: In double-blind period, participants received placebo matched to guselkumab (400 milligrams [mg]) intravenous (IV) infusion at Weeks 0, 4 and 8 and placebo matched to guselkumab (200 mg) subcutaneous (SC) injection every 4 weeks (q4w) from Week 12 through Week 48 along with standard-of-care treatment of mycophenolate mofetil (MMF)/mycophenolic acid (MPA) and glucocorticoids. Participants who achieved complete renal response (CRR) at Week 48 and 52, and completed the Week 52 assessments entered the long-term extension (LTE) phase and continued to receive placebo matched to guselkumab SC injection q4w from Week 52 through Week 84 (that is., up to LTE phase treatment termination).
- Guselkumab: In double-blind period, participants received guselkumab 400 mg IV infusion at Weeks 0, 4, and 8 and guselkumab 200 mg SC injection q4w from Week 12 through Week 48 along with standard-of-care treatment of MMF/MPA and glucocorticoids. Participants who achieved CRR at Week 48 and 52, and completed the Week 52 assessments entered LTE phase and continued to receive guselkumab 200 mg SC injection q4w from Week 52 through Week 84 (that is., up to LTE phase treatment termination).
Period: Double Blind Period: Week 0 to Week 52
Arm/Group | Placebo | Guselkumab
Started | 16 | 17
Completed | 9 | 8
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study Terminated by Sponsor | 6 | 8
Period: LTE Phase:Week 52 to 96(LTE Termination)
Arm/Group | Placebo | Guselkumab
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Protocol-specified withdrawal criterion met | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study Terminated by Sponsor | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (11.69) | 35.3 (10.07) | 37 (10.86)
Age, Customized [Count of Participants; unit: Participants]
  >= 55 years | 1 | 1 | 2
  < 55 years | 15 | 16 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 14 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 5 | 4 | 9
  MEXICO | 1 | 3 | 4
  RUSSIAN FEDERATION | 2 | 1 | 3
  TAIWAN | 3 | 0 | 3
  THAILAND | 0 | 1 | 1
  UKRAINE | 5 | 7 | 12
  UNITED STATES | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least 50 Percent (%) Decrease From Baseline in Proteinuria at Week 24
Description: Percentage of participants achieving at least 50% decrease in proteinuria from baseline at Week 24 was reported. Proteinuria analysis was based on urine protein creatinine ratio (UPCR) and was defined as the presence of an excess of serum proteins in the urine, which may be an early sign of kidney disease.
Time Frame: Week 24
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
percentage of participants | 56.3 | 35.3

2. Secondary Outcome: Percentage of Participants Who Achieved Complete Renal Response (CRR) at Week 24
Description: Percentage of participants who achieved CRR at Week 24 were reported. CRR was defined as UPCR less than (<) 0.5 milligrams per milligrams (mg/mg), estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 60 milliliter per minute per 1.73 meter square (mL/min/1.73m^2) or no confirmed decrease >=20% from baseline and prednisone dose less than or equal to (<=) 10 milligrams per day (mg/d). Participant was considered as achieved CRR who did not discontinue study intervention for any reason excluding COVID-19 related discontinuations or met the medication intercurrent event (exceeded baseline glucocorticoid dose, increase above 10 mg/d prednisone equivalent after Week 12, use of new or increased dose of concomitant medication related to LN or other immunosuppressive agents, within 8 weeks prior to the outcome measure (OM) time point (Week 24) or initiation of prohibited medications at any time prior to the endpoint time point (Week 24).
Time Frame: Week 24
Population: FAS included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
percentage of participants | 18.8 | 17.6

3. Secondary Outcome: Percentage of Participants Who Achieved CRR at Week 52
Description: Percentage of participants who achieved CRR at Week 52 were reported. CRR was defined as UPCR less than (<) 0.5 mg/mg, eGFR >= 60 mL/min/1.73m^2 or no confirmed decrease >=20% from baseline and prednisone dose <= 10 mg/d. Participant was considered as achieved CRR who did not discontinue study intervention for any reason excluding COVID-19 related discontinuations or met the medication intercurrent event (exceeded baseline glucocorticoid dose, increase above 10 mg/d prednisone equivalent after Week 12, use of new or increased dose of concomitant medication related to LN or other immunosuppressive agents, within 8 weeks prior to the outcome measure time point (Week 52) or initiation of prohibited medications at any time prior to the outcome measure time point (Week 52).
Time Frame: Week 52
Population: The Full Analyses Set for Week 52 (FASC52) included all randomized participants who received at least 1 dose of any study intervention and had the opportunity to complete the Week 52 visit prior to study termination. Here 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 12 | 11
percentage of participants | 25.0 | 9.1

4. Secondary Outcome: Percentage of Participants Achieving a Sustained Reduction in Steroid Dose <=10 mg/d of Prednisone or Equivalent From Week 16 Through Week 24
Description: Percentage of participants achieving a sustained reduction in steroid dose less than or equal to (<=) 10 mg/day of prednisone or equivalent from week 16 through Week 24were reported.
Time Frame: From Week 16 through Week 24
Population: FAS included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
percentage of participants | 87.5 | 94.1

5. Secondary Outcome: Percentage of Participants Achieving at Least 50% Decrease in Proteinuria From Baseline at Week 52
Description: Percentage of participants achieving at least 50% decrease in proteinuria from baseline at Week 52 were reported. Proteinuria analysis was based on urine protein creatinine ratio (UPCR) and was defined as the presence of an excess of serum proteins in the urine, which may be an early sign of kidney disease.
Time Frame: Week 52
Population: FASC52 included all randomized participants who received at least 1 dose of any study intervention and had the opportunity to complete the Week 52 visit prior to study termination. Here 'N' (number of participants analysed) signifies participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 12 | 11
percentage of participants | 25.0 | 27.3

6. Secondary Outcome: Percentage of Participants With Urine Protein to Creatinine Ratio (UPCR) < 0.5 mg/mg at Week 24
Description: Percentage of participants with UPCR <0.5 mg/mg at Week 24 were reported.
Time Frame: Week 24
Population: FAS included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
percentage of participants | 25.0 | 29.4

7. Secondary Outcome: Percentage of Participants With UPCR < 0.75 mg/mg at Week 24
Description: Percentage of participants with UPCR less than 0.75 mg/mg at Week 24 were reported.
Time Frame: Week 24
Population: FAS included all randomized participants who received at least 1 dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
percentage of participants | 37.5 | 35.3

8. Secondary Outcome: Percentage of Participants Who Achieved CRR Through Week 24
Description: Percentage of participants who achieved CRR through Week 24 was reported. CRR was defined as UPCR<0.5 mg/mg, eGFR >= 60 mL/min/1.73m^2 or no confirmed decrease>=20% from baseline and prednisone dose <= 10 mg/d. Participant was considered as achieved CRR who did not discontinue study intervention for any reason excluding COVID-19 related discontinuations or met the medication intercurrent event (exceeded baseline glucocorticoid dose, increase above 10 mg/d prednisone equivalent after Week 12, use of new or increased dose of concomitant medication related to lupus nephritis (LN) or other immunosuppressive agents, within 8 weeks prior to the outcome measure time point (Week 24) or initiation of prohibited medications at any time prior to the outcome measure time point (Week 24).
Time Frame: Up to Week 24
Population: FAS included all randomized participants who received at least 1 dose of any study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Percentage of participants | 37.5 | 23.5
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p = 0.7807, log-rank test; Hazard Ratio (HR) = 0.62, 80% CI 2-sided [0.27 to 1.41] — Hazard ratio and 80% CI: estimated by Cox proportional hazards model adjusting for baseline UPCR level (<3 mg/mg and >=3 mg/mg)

9. Secondary Outcome: Percentage of Participants With Treatment Failure (TF) Through Week 52
Description: Percentage of participants with TF through Week 52 was reported. TF was defined as time to the first occurrence of TF from baseline. Participant was considered to have treatment failure, who did not continue study intervention for any reason excluding COVID-19 related discontinuations or met the medication intercurrent event (exceeded baseline glucocorticoid dose, increase above 10 mg/d prednisone equivalent after Week 12, use of new or increased dose of concomitant medication related to LN or other immunosuppressive agents, within 8 weeks prior to the outcome measure time point (Week 52) or initiation of prohibited medications at any time prior to the outcome measure time point (Week 52).
Time Frame: Up to Week 52
Population: FAS included all randomized participants who received at least 1 dose of any study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Percentage of participants | 18.8 | 35.3
Statistical Analysis 1: Comparison: Placebo vs Guselkumab; Test type: Superiority; p = 0.4654, long-rank test; Hazard Ratio (HR) = 1.52, 80% CI 2-sided [0.62 to 3.85] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with AEs were reported. An AE was defined as any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product did not necessarily have a causal relationship with the treatment. Therefore, it could be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.
Time Frame: DB period: From Week 0 up to 12 week safety follow-up (i.e., up to Week 60); LTE phase: From Week 52 up to LTE phase termination (i.e., up to Week 96)
Population: Safety analysis set (SAS) included all participants who received at least one dose of study intervention. Since a small number of participants only entered the LTE phase than the planned enrollment count, no separate adverse events analysis was performed for the LTE phase participants and thus, data of both DB period and LTE phase were presented together for this outcome measure under the arms: placebo and guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 12 | 12

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of Participants with SAEs were reported. An AE was defined as any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product did not necessarily have a causal relationship with the treatment. Therefore, it could be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. A SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product, or was medically important.
Time Frame: as for outcome 10
Population: SAS included all participants who received at least one dose of study intervention. Since a small number of participants only entered the LTE phase than the planned enrollment count, no separate adverse events analysis was performed for the LTE phase participants and thus, data of both DB period and LTE phase were presented together for this outcome measure under the arms: placebo and guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 1 | 1

12. Secondary Outcome: Number of Participants With Related AEs
Description: Number of participants with related AEs were reported. An AE was defined as any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product did not necessarily have a causal relationship with the treatment. Therefore, it could be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. Related AE was defined as the AE assessed by the investigator related to study agent.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 2 | 2

13. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation of Study Intervention
Description: Number of participants with AEs leading to discontinuation of study intervention were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 1 | 2

14. Secondary Outcome: Number of Participants With Infections
Description: Number of participants with infections as assessed by the investigator were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 5 | 6

15. Secondary Outcome: Number of Participants With Serious Infections
Description: Number of participants with serious infections as assessed by the investigator were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Infections Requiring Oral or Parenteral Antimicrobial Treatment
Description: Number of participants with infections requiring oral or parenteral antimicrobial treatment planned to be were reported.
Time Frame: as for outcome 10
Population: SAS included all participants who received at least one dose of study intervention. For this outcome measure, no data was collected and analyzed due to premature termination of the study.
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants With AEs Temporally Associated With an Infusion
Description: Number of participants with AEs temporally (a reaction that occurred during or within 1 hour after infusion) associated with an infusion were reported. AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product does not necessarily have a causal relationship with the treatment. Therefore, it can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 1 | 0

18. Secondary Outcome: Number of Participants With AEs With Injection-site Reactions
Description: Number of participants with injection-site reactions as assessed by the investigator were reported. An injection-site reaction is any adverse reaction at a SC study intervention injection-site.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants | 1 | 0

19. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Activated Partial Thromboplastin Time
Description: Change from baseline in clinical laboratory parameter: activated partial thromboplastin time was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS included all participants who received at least one dose of study intervention. Here 'n' (number analyzed) signifies the number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies number of participants with available data for this OM. Since a small number of participants only entered LTE phase than planned enrollment count, planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this OM.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 12 | 13
Seconds
  Week 24 | 0.78 (1.734) | 0.96 (3.869)
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | 0.88 (1.387) |

20. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Basophils
Description: Change from baseline in clinical laboratory parameter: basophils was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS included all subjects who received at least one dose of study intervention. Here 'n' (number analyzed) signifies number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies to number of participants with available data for this OM. Since a small number of participants only entered LTE phase than planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this OM.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^9 cells per liter
  Week 24 | -0.009 (0.0512) | -0.009 (0.0502)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -0.070 (0.0990) |

21. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Eosinophils
Description: Change from baseline in clinical laboratory parameter: eosinophils was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS population. Here 'n' (number analyzed) signifies the number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^9 cells per liter
  Week 24 | 0.022 (0.0472) | -0.041 (0.1620)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | 0.000 (0.0283) |

22. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Change from baseline in clinical laboratory parameter: erythrocytes mean corpuscular hemoglobin was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: petagram (pg)
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
petagram (pg)
  Week 24 | 0.1 (1.38) | -0.8 (1.06)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -1.5 (2.12) |

23. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Erythrocytes Mean Corpuscular Volume
Description: Change from baseline in clinical laboratory parameter: erythrocytes mean corpuscular volume was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 11
femtoliter (fL)
  Week 24 | 0.5 (6.35) | -3.3 (5.37)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -4.0 (0.00) |

24. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Erythrocytes
Description: Change from baseline in clinical laboratory parameter: erythrocytes was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS included all subjects who received at least one dose of study intervention. Here 'n' (number analyzed) signifies number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants with available data for this OM. Since a small number of participants only entered the LTE phase than planned enrollment count, planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this OM.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^12 cells per liter
  Week 24 | -0.16 (0.582) | 0.12 (0.577)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -0.40 (0.566) |

25. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Hematocrit
Description: Change from baseline in clinical Laboratory parameter: hematocrit was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS included all participants who received at least one dose of study intervention. Here 'n' refers to the number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants with available data for this OM. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this OM.
Measure: Mean (Standard Deviation); unit: percentage of blood cells
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 11
percentage of blood cells
  Week 24 | -0.013 (0.0411) | -0.004 (0.0356)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -0.055 (0.0495) |

26. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Hemoglobin
Description: Change from baseline in clinical laboratory parameter: hemoglobin was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
grams per liter (g/L)
  Week 24 | -5.2 (15.57) | -0.3 (14.82)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -17.0 (22.63) |

27. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter Leukocytes
Description: Change from baseline in clinical laboratory parameter: leukocytes was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS population. Here 'n' (number analyzed) signifies the number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants of both with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^9 cells per liter
  Week 24 | -0.622 (3.8729) | -1.157 (3.1246)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -5.120 (7.7499) |

28. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Lymphocytes
Description: Change from baseline in clinical laboratory parameter: lymphocytes was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS population. Here 'n' (number analyzed) signifies to number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants of both with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^9 cells per Liter
  Week 24 | 0.006 (0.5213) | -0.032 (0.3860)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -0.545 (1.0960) |

29. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Monocytes
Description: Change from baseline in clinical laboratory parameter: monocytes was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS population. Here 'n' (number analyzed) signifies to the number of participants evaluable at specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^9 cells per liter
  Week 24 | -0.014 (0.3277) | -0.002 (0.1268)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -0.510 (0.7354) |

30. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Hematology Parameter: Segmented Neutrophils
Description: Change from baseline in clinical laboratory parameter: segmented neutrophils was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^9 cells per liter
  Week 24 | -0.630 (3.2494) | -1.074 (2.9652)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -3.990 (5.8548) |

31. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Platelets
Description: Change from baseline in clinical laboratory parameter: platelets was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
10^9 cells per liter
  Week 24 | -36.7 (61.43) | -17.8 (61.89)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -70.5 (67.18) |

32. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Prothrombin International Normalized Ratio
Description: Change from baseline in clinical laboratory parameter: prothrombin international normalized ratio was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 13
Ratio
  Week 24 | 0.02 (0.090) | 0.01 (0.064)
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | 0.00 (0.000) |

33. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Prothrombin Time
Description: Change from baseline in clinical laboratory parameter: prothrombin time was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 13
second
  Week 24 | 0.18 (0.766) | 0.16 (0.425)
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | -0.03 (0.359) |

34. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Reticulocytes/Erythrocytes
Description: Change from baseline in clinical laboratory hematology parameter:reticulocytes/erythrocytes was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: percentage of blood cells
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 11
percentage of blood cells
  Week 24 | -0.0007 (0.00485) | -0.0001 (0.00541)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | 0.0000 (0.01414) |

35. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Alanine Aminotransferase
Description: Change from baseline in clinical laboratory parameter: alanine aminotransferase was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Enzyme units per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
Enzyme units per liter
  Week 24 | 2.6 (10.98) | -3.1 (6.57)
  Week 52: number analyzed (Participants) | 4 | 0
  Week 52 | 2.3 (4.92) |

36. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Albumin
Description: Change from baseline in clinical laboratory parameter: albumin was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
Grams per Liter (g/L)
  Week 24 | 2.4 (5.57) | 1.9 (4.58)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 3.5 (5.32) | -3.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

37. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Alkaline Phosphatase
Description: Change from baseline in clinical laboratory parameter: alkaline phosphatase was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Enzyme units per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
Enzyme units per liter
  Week 24 | 1.9 (16.75) | 1.7 (8.07)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 6.5 (5.00) | 6.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

38. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Aspartate Aminotransferase
Description: Change from baseline in clinical laboratory parameter: aspartate aminotransferase was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Enzyme units per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 13
Enzyme units per liter
  Week 24 | 0.0 (4.97) | -0.7 (5.41)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 1.5 (2.38) | 1.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

39. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Bicarbonate
Description: Change from baseline in clinical laboratory parameter: bicarbonate was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: SAS population. Here 'n' (number analyzed) signifies the number of participants evaluable at specified timepoints. Here 'N' number of participants analyzed) signifies the number of participants with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 13 | 12
mmol/L
  Week 24 | -0.78 (4.97) | 0.21 (5.41)
  Week 52: number analyzed (Participants) | 2 | 0
  Week 52 | -2.20 (2.38) |

40. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Bilirubin
Description: Change from baseline in clinical laboratory parameter: bilirubin was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
micromole per liter
  Week 24 | 0.1 (1.98) | 0.3 (2.46)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | -0.3 (2.06) | 4.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

41. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: Calcium
Description: Change from baseline in clinical laboratory parameter: calcium was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
mmol/L
  Week 24 | 0.039 (0.1172) | 0.073 (0.0958)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 0.000 (0.1871) | 0.010 (NA) — Here, NA signifies that SD could not be calculated for single participant.

42. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Chloride
Description: Change from baseline in clinical laboratory parameter: chloride was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
mmol/L
  Week 24 | 0.1 (4.50) | 0.7 (0.0958)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 2.0 (4.83) | 2.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

43. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: Cholesterol
Description: Change from baseline in clinical laboratory parameter: cholesterol was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 15
mmol/L
  Week 24 | -1.325 (1.3026) | 0.017 (0.7818)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | -2.235 (1.6588) | 0.210 (NA) — Here, NA signifies that SD could not be calculated for single participant.

44. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Creatine Kinase
Description: Change from baseline in clinical laboratory parameter: creatine kinase was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Enzyme units per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
Enzyme units per liter
  Week 24 | 3.3 (42.22) | -0.5 (53.94)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | -8.8 (36.65) | -2.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

45. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Creatinine
Description: Change from baseline in clinical laboratory parameter: creatinine was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
micromole per liter
  Week 24 | 0.6 (18.30) | 6.7 (16.78)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | -3.3 (7.54) | -5.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

46. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Protein
Description: Change from baseline in clinical laboratory parameter: protein was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
g/L
  Week 24 | 3.0 (8.83) | 2.9 (16.78)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 7.0 (7.39) | 1.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

47. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Phosphate
Description: Change from baseline in clinical laboratory parameter: phosphate was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
mmol/L
  Week 24 | 0.060 (0.1498) | 0.030 (0.2916)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | -0.035 (0.2213) | 0.220 (NA) — Here, NA signifies that SD could not be calculated for single participant.

48. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Sodium
Description: Change from baseline in clinical laboratory parameter: sodium was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
mmol/L
  Week 24 | -0.7 (2.30) | 0.4 (4.24)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 1.0 (1.41) | 3.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

49. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: Potassium
Description: Change from baseline in clinical laboratory parameter: potassium was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
mmol/L
  Week 24 | 0.19 (0.704) | 0.13 (0.402)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 0.03 (0.457) | 0.00 (NA) — Here, NA signifies that SD could not be calculated for single participant.

50. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameters: Urea Nitrogen
Description: Change from baseline in clinical laboratory parameter: urea nitrogen was reported.
Time Frame: Baseline (Week 0), Week 24, and Week 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
mmol/L
  Week 24 | -1.23 (3.106) | 0.71 (2.177)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | -1.60 (1.564) | 0.50 (NA) — Here, NA signifies that SD could not be calculated for single participant.

51. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Glomerular Filtration Rate (GFR) From Creatinine Adjusted for Body Surface Area (BSA)
Description: Change from baseline in clinical laboratory parameter: GFR from Creatinine Adjusted for BSA was reported.
Time Frame: Baseline (Week 0), Weeks 24 and 52
Population: SAS population. Here 'n' (number analyzed) refers to the number of participants evaluable at each specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants of both with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: milliliter/minute/1.73 meter square
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
milliliter/minute/1.73 meter square
  Week 24 | 0.44 (21.639) | -5.87 (17.150)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 6.75 (22.588) | 5.60 (NA) — Here, NA signifies that SD could not be calculated for single participant.

52. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Gamma Glutamyl and Transferase Lactate Dehydrogenase
Description: Change from baseline in clinical laboratory parameter: gamma glutamyl transferase and lactate dehydrogenase were reported.
Time Frame: Baseline (Week 0), Weeks 24 and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: Enzyme units per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
Enzyme units per liter
  gamma glutamyl transferase: Week 24 | -0.6 (15.01) | -3.0 (9.70)
  gamma glutamyl transferase: Week 52: number analyzed (Participants) | 4 | 1
  gamma glutamyl transferase: Week 52 | 1.0 (8.60) | -2.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.
  Lactate dehydogenase: Week 24: number analyzed (Participants) | 13 | 12
  Lactate dehydogenase: Week 24 | -14.5 (47.90) | -2.5 (17.52)
  Lactate dehydogenase: Week 52: number analyzed (Participants) | 2 | 1
  Lactate dehydogenase: Week 52 | -62.5 (40.31) | 7.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

53. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Glucose and Magnesium
Description: Change from baseline in clinical laboratory parameter: glucose and magnesium were reported.
Time Frame: Baseline, Weeks 24, 52
Population: SAS population. Here 'n' (number analyzed) signifies the number of participants evaluable at each specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants of both with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
millimoles per liter (mmol/L)
  Glucose: Week 24 | -0.23 (1.041) | -0.04 (0.908)
  Glucose:: Week 52: number analyzed (Participants) | 4 | 1
  Glucose:: Week 52 | -0.03 (0.126) | 0.20 (NA) — Here, NA signifies that SD could not be calculated for single participant.
  Magnesium: Week 24 | -0.024 (0.0696) | -0.022 (0.0607)
  Magnesium: Week 52 | -0.068 (0.0842) | -0.010 (NA) — Here, NA signifies that SD could not be calculated for single participant.

54. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Protein
Description: Change from baseline in clinical laboratory parameter: protein was reported.
Time Frame: Baseline (Week 0), Weeks 24 and 52
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
gram per Liter (g/L)
  Week 24 | 3.0 (8.83) | 2.9 (6.55)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | 7.0 (7.39) | 1.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

55. Secondary Outcome: Change From Baseline in Chemistry Parameters: Protein/Creatinine
Description: Change from baseline in chemistry parameter: protein/creatinine was reported.
Time Frame: Baseline, Weeks 24 and 52
Population: SAS population. Here 'n' (number analyzed) signifies the number of participants evaluable at each specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 15 | 16
mg/mg
  Week 24: number analyzed (Participants) | 14 | 16
  Week 24 | -1.509 (1.9494) | -0.821 (2.4250)
  Week 52: number analyzed (Participants) | 4 | 7
  Week 52 | -1.586 (1.7966) | -0.352 (1.6960)

56. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Urate
Description: Change from baseline in clinical laboratory parameter: urate was reported.
Time Frame: Baseline, Weeks 24, 52
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 14 | 16
micromole per liter
  Week 24 | -73.4 (104.11) | 8.4 (48.61)
  Week 52: number analyzed (Participants) | 4 | 1
  Week 52 | -79.5 (79.38) | -2.0 (NA) — Here, NA signifies that SD could not be calculated for single participant.

57. Secondary Outcome: Change From Baseline in Clinical Laboratory Parameter: Urine Protein
Description: Change from baseline in clinical laboratory parameter: urine protein was reported.
Time Frame: Baseline (Week 0), Weeks 24 and 52
Population: SAS population.Here 'n' (number analyzed) signifies the number of participants evaluable at each specified timepoints. Here 'N' (number of participants analyzed) signifies the number of participants of both with available data for this outcome measure. Since a small number of participants only entered the LTE phase than the planned enrollment count, the planned analysis of change from baseline for the safety parameters was not performed for the LTE phase for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram per liter
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 15 | 17
milligram per liter
  Week 24: number analyzed (Participants) | 15 | 16
  Week 24 | -1322.1 (1865.82) | -310.3 (1494.58)
  Week 52: number analyzed (Participants) | 6 | 7
  Week 52 | -1821.7 (2334.78) | -166.4 (1099.54)

58. Secondary Outcome: Number of Participants With Maximum US National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Toxicity Grade (Grade 4) in Clinical Laboratory Parameters: Hematology and Chemistry
Description: Number of participants with maximum US NCI-CTCAE toxicity grade (Grade 4) in clinical laboratory parameters: hematology and chemistry were reported. Toxicity were graded as Grade 1: Mild, Grade 2: Moderate; Grade 3: Severe. Grade 4: Life-threatening and Grade 5: Death.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
Participants
  Alanine Aminotransferase Increased | 0 | 0
  Alkaline Phosphatase Increased | 0 | 0
  Aspartate Aminotransferase Increased | 0 | 0
  Blood Bilirubin Increased | 0 | 0
  CPK Increased | 0 | 0
  Cholesterol High | 0 | 0
  Creatinine Increase | 0 | 0
  GGT Increased | 0 | 0
  Hypermagnesemia | 0 | 0
  Hypernatremia | 0 | 0
  Hypertriglyceridemia | 0 | 0
  Hypoalbuminemia | 0 | 0
  Hypoglycemia | 0 | 0
  Hypokalemia | 0 | 0
  Hypomagnesemia | 0 | 0
  Hyponatremia | 0 | 0
  Activated Partial Thromboplastin Time Prolonged | 0 | 0
  Anemia | 0 | 0
  Hemoglobin Increased | 0 | 0
  Leukocytosis | 0 | 0
  Lymphocyte Count Decreased | 0 | 0
  Lymphocyte Count Increased | 0 | 0
  Neutrophil Count Decreased | 0 | 0
  Platelet Count Decreased | 0 | 0
  White Blood Cell Decreased | 0 | 0

59. Secondary Outcome: Percentage of Participants With Abnormal Vital Signs: Systolic and Diastolic Blood Pressure
Description: Percentage of participants with abnormal vital signs: Systolic and Diastolic blood pressure were reported.
Time Frame: Up to Week 60
Population: SAS included all participants who received at least one dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab
Number analyzed (Participants) | 16 | 17
percentage of participants
  Systolic Blood Pressure: <85 mmHg | 0 | 0
  Systolic Blood Pressure::>180 mmHg | 6.3 | 5.9
  Diastolic Blood Pressure: <55 mmHg | 6.3 | 0
  Diastolic Blood Pressure: >115 mmHg | 6.3 | 0

60. Secondary Outcome: Serum Concentration of Guselkumab
Description: Serum Concentration of guselkumab were reported.
Time Frame: Predose: Weeks 0,4,8,12,16,20,24, 36; Post-dose: Week 0 (1 hour after intravenous administration), Day 2, Week 52 and 60
Population: Pharmacokinetic analysis set included all participants who received at least 1 administration of guselkumab and had at least one post-dose sample collection. Here 'n' (number analyzed) signifies number of participants evaluable at specified timepoints. Data for this OM was not planned to be collected and analyzed for placebo arm. Since small number of participants only entered LTE phase than the planned enrollment, planned serum concentration analysis was not performed for LTE phase for this OM.
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Guselkumab
Number analyzed (Participants) | 16
microgram/milliliter
  Week 0, predose | 0.00 (0.000)
  Week 0, 1h after IV administration | 146.20 (41.273)
  Day 2, post-dose | 96.55 (33.805)
  Week 4, predose | 11.20 (7.175)
  Week 8, predose: number analyzed (Participants) | 15
  Week 8, predose | 12.85 (9.549)
  Week 12, predose: number analyzed (Participants) | 14
  Week 12, predose | 18.17 (11.784)
  Week 16, pre-dose: number analyzed (Participants) | 13
  Week 16, pre-dose | 9.89 (5.016)
  Week 20, predose: number analyzed (Participants) | 14
  Week 20, predose | 7.63 (4.689)
  Week 24, predose: number analyzed (Participants) | 12
  Week 24, predose | 6.42 (3.447)
  Week 36, predose: number analyzed (Participants) | 10
  Week 36, predose | 6.57 (1.827)
  Week 52, post-dose: number analyzed (Participants) | 6
  Week 52, post-dose | 6.13 (3.262)
  Week 60, post-dose: number analyzed (Participants) | 4
  Week 60, post-dose | 0.39 (0.641)

61. Secondary Outcome: Number of Participants With Treatment-boosted Anti-drug Antibodies (ADA) Response
Description: Treatment-boosted ADA positive participants: participants who were positive at baseline and whose titers increased 2-fold at any time after treatment. Titer values were categorized as<=1:10, 10 to 100, 100 to 1000, >1000.
Time Frame: From Baseline (Week 0) through Week 24 and Week 60
Population: Immunogenecity analysis set inlcuded all participants who received at least 1 administration of guselkumab and had at least one post-dose sample collection. Here 'n' (number analyzed) signifies the number of participants evaluable at specified timepoints. Data for this outcome measure was not planned to be collected and analyzed for the placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab
Number analyzed (Participants) | 17
Participants
  Week 24 | 1
  Week 60: number analyzed (Participants) | 16
  Week 60 | 1

ADVERSE EVENTS:
Time Frame: DB period: From Week 0 up to 12 week safety follow-up (i.e., up to Week 60); LTE phase: From Week 52 up to LTE phase termination (i.e., up to Week 96)
Description: SAS included all participants who received at least one dose of study intervention. Since a small number of participants only entered the LTE period than the planned enrollment count, no separate adverse events analysis was performed for the LTE phase participants and thus, data of both DB period and LTE phase were presented together for AEs (SAEs and non- SAEs) and all cause mortality data under the arms: placebo and guselkumab.
Arm/Group | Placebo | Guselkumab
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/17
Other Adverse Events (participants affected / at risk) | 12/16 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Guselkumab (N=17)
Basal Ganglia Stroke (Nervous system disorders) | 1 | 0
Lupus Nephritis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Guselkumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Ocular Myasthenia (Eye disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Chronic Gastritis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Injection Site Erythema (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 0 | 2
Pneumonia Bacterial (Infections and infestations) | 1 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 2
Medication Error (Injury, poisoning and procedural complications) | 0 | 2
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Blood Bicarbonate Decreased (Investigations) | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1
Heart Rate Increased (Investigations) | 0 | 1
Liver Function Test Increased (Investigations) | 0 | 1
White Blood Cell Count Increased (Investigations) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Sle Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Tension Headache (Nervous system disorders) | 1 | 0
Lupus Nephritis (Renal and urinary disorders) | 2 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Striae (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to enrollment challenges, the Sponsor decided to stop screening of new participants and stop the study early. Since a small number of participants only entered the LTE phase than the planned enrollment count, some of the planned safety analyses were not performed for the LTE phase participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT04376827/Prot_002.pdf
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT04376827/SAP_003.pdf